CLINICAL TRIAL: NCT04987333
Title: A Phase 1, Open-label, Sequential-group, Single-dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of AMG 592 Administered Subcutaneously in Healthy Chinese, Japanese, and Caucasian Subjects
Brief Title: Study of Efavaleukin Alfa in Healthy Chinese, Japanese, and Caucasian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20200102
Record Dates: First submitted 2021-07-26; First posted 2021-08-03 (Actual); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2023-10

CONDITIONS: Inflammatory Diseases
Keywords: Systemic lupus erythematosus (SLE); Steroid-refractory chronic graft-versus-host disease (GvHD); Ulcerative colitis; Single-dose study; Efavaleukin alfa; Regulatory T Cells (Tregs); Inflammatory
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Colitis, Ulcerative

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group 1: Chinese participants - efavaleukin alfa dose level 1 (Experimental): Chinese participants will receive a single dose of efavaleukin alfa at dose level 1.
  Interventions: Drug: Efavaleukin alfa
- Group 2: Chinese participants - efavaleukin alfa dose level 2 (Experimental): Chinese participants will receive a single dose of efavaleukin alfa at dose level 2.
  Interventions: Drug: Efavaleukin alfa
- Group 3: Japanese participants - efavaleukin alfa dose level 2 (Experimental): Japanese participants will receive a single dose of efavaleukin alfa at dose level 2.
  Interventions: Drug: Efavaleukin alfa
- Group 4: Caucasian participants - efavaleukin alfa dose level 2 (Experimental): Caucasian participants will receive a single dose of efavaleukin alfa at dose level 2.
  Interventions: Drug: Efavaleukin alfa

INTERVENTIONS:
Drug: Efavaleukin alfa — Administered as a single dose SC injection.

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetics (PK) of efavaleukin alfa after single subcutaneous (SC) administration in healthy Chinese, Japanese, and Caucasian participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female participants, between 18 and 55 years of age (inclusive) at the time of Screening.
* Chinese, Japanese, or Caucasian participant:

  * Chinese participants must be of Chinese ancestry (4 grandparents and biological parents).
  * Japanese participants must be first- or second-generation Japanese (4 grandparents and biological parents; participant or both of their parents must have been born in Japan).
  * Caucasian participants are those who self-identify exclusively as such on the electronic case report form (eCRF) and also identify their biological parents as such.
* In good health, determined by no clinically significant findings from medical history, physical examinations, 12-lead electrocardiogram (ECG), vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) as assessed by the Investigator (or designee).
* Body mass index between 17 and 30 kg/m^2 (inclusive) at the time of Screening.

Exclusion Criteria:

* Evidence of scars, tattoos, or other skin lesions that may interfere with the injection site or injection site assessments.
* History or evidence of clinically significant arrhythmia at Screening, including any clinically significant findings on the ECG taken at Check-in.
* A QT interval corrected for heart rate using Fridericia's method (QTcF) interval > 450 msec in male participants or > 470 msec in female participants or history/evidence of long QT syndrome, at Screening or Check-in.
* PR interval > 210 msec, at Screening or Check-in.
* Second- or third-degree atrioventricular (AV) block , at Screening or Check-in.
* Systolic blood pressure (BP) > 140 mmHg or < 90 mmHg, or diastolic BP > 90 mmHg, or HR > 100 bpm, at Screening or Check-in.
* Estimated glomerular filtration rate less than 60 mL/min/1.73 m^2 as calculated by the Modification of Diet in Renal Disease equation, at Screening.
* HbA1C ≥ 7%, at Screening or Check-in.
* Participants who have received live vaccines within 5 weeks prior to Screening, or plan to receive live vaccines within 105 days after administration of an investigational product.
* Positive hepatitis B or hepatitis C panel (ie, positive hepatitis B surface antigen, hepatitis B core antibody or hepatitis C antibody) at Screening, or a medical history for hepatitis B or C; and/or positive human immunodeficiency virus test, at Screening. Participants whose results are compatible with prior vaccination may be included. Participants with a history of hepatitis B vaccination without a history of hepatitis B or C are allowed to participate.
* Consumption of foods and beverages containing poppy seeds within 7 days prior to Check-in.
* History of alcoholism or drug/chemical abuse within 1 year prior to Check-in.
* Use of tobacco- or nicotine-containing products within 6 months prior to Check-in.
* Positive test for illicit drugs, cotinine (tobacco or nicotine use), and/or alcohol use at Screening or Check-in.
* Female participants with a positive pregnancy test at Screening or Check-in.
* Participant has received a dose of an investigational drug within the past 90 days or 5 half-lives of the drug, whichever is longer, prior to Check-in.
* Donation of blood from 90 days prior to Check-in, plasma from 2 weeks prior to Check-in, or platelets from 6 weeks prior to Check-in.
* Participants with abnormal laboratory results for alanine aminotransferase (ALT) or aspartate aminotransferase (AST) (ie, > upper limit of normal) and total bilirubin (ie, > upper limit of normal) at Screening and Check-in.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Labcorp Clinical Research Unit - Leeds, Leeds, LDS, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 1 research center in the United Kingdom from August 2021 to October 2022.
Groups:
- Group 1: Chinese Participants - Efavaleukin Alfa (Dose Level 1): Chinese participants who received efavaleukin alfa administered as one subcutaneous (SC) injection at dose level 1 (low).
- Group 2: Chinese Participants - Efavaleukin Alfa (Dose Level 2): Chinese participants who received efavaleukin alfa administered as one SC injection at dose level 2 (high).
- Group 3: Japanese Participants -Efavaleukin Alfa (Dose Level 2): Japanese participants who received efavaleukin alfa administered as one SC injection at dose level 2 (high).
- Group 4: Caucasian Participants - Efavaleukin Alfa (Dose Level 2): Caucasian participants who received efavaleukin alfa administered as one SC injection at dose level 2 (high).
Period: Overall Study
Arm/Group | Group 1: Chinese Participants - Efavaleukin Alfa (Dose Level 1) | Group 2: Chinese Participants - Efavaleukin Alfa (Dose Level 2) | Group 3: Japanese Participants -Efavaleukin Alfa (Dose Level 2) | Group 4: Caucasian Participants - Efavaleukin Alfa (Dose Level 2)
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who received at least 1 dose of efavaleukin alfa and had at least 1 postdose safety assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Chinese Participants - Efavaleukin Alfa (Dose Level 1) | Group 2: Chinese Participants - Efavaleukin Alfa (Dose Level 2) | Group 3: Japanese Participants -Efavaleukin Alfa (Dose Level 2) | Group 4: Caucasian Participants - Efavaleukin Alfa (Dose Level 2) | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.9 (4.55) | 28.3 (4.86) | 29.5 (4.11) | 37.9 (12.01) | 30.9 (7.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 2 | 5 | 15
  Male | 5 | 3 | 6 | 3 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 8 | 8 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8 | 8 | 8 | 0 | 24
  White | 0 | 0 | 0 | 8 | 8

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Efavaleukin Alfa
Description: Blood samples were collected to determine PK parameters.
Time Frame: Day 1: Pre-dose, 6, 12, & 16 hours post-dose, and days 2 (24 hours post-dose), 3, 4, 5, 6, 8, 11, 15, 22, 29 and 43
Population: Pharmacokinetic (PK) population: all participants who received at least 1 dose of efavaleukin alfa and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group 1: Chinese Participants - Efavaleukin Alfa (Dose Level 1) | Group 2: Chinese Participants - Efavaleukin Alfa (Dose Level 2) | Group 3: Japanese Participants -Efavaleukin Alfa (Dose Level 2) | Group 4: Caucasian Participants - Efavaleukin Alfa (Dose Level 2)
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng/mL | 26.9 (52.1) | 41.6 (33.4) | 48.1 (33.0) | 56.1 (47.7)

2. Primary Outcome: Time of the Maximum Observed Serum Concentration (Tmax) of Efavaleukin Alfa
Description: Blood samples were collected to determine PK parameters.
Time Frame: Day 1: Pre-dose, 6, 12, & 16 hours post-dose, and days 2 (24 hours post-dose), 3, 4, 5, 6, 8, 11, 15, 22, 29 and 43
Population: PK population: all participants who received at least 1 dose of efavaleukin alfa and had evaluable PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1: Chinese Participants - Efavaleukin Alfa (Dose Level 1) | Group 2: Chinese Participants - Efavaleukin Alfa (Dose Level 2) | Group 3: Japanese Participants -Efavaleukin Alfa (Dose Level 2) | Group 4: Caucasian Participants - Efavaleukin Alfa (Dose Level 2)
Number analyzed (Participants) | 8 | 8 | 8 | 8
hours | 24.0 [24.0 to 48.1] | 24.0 [16.0 to 48.0] | 24.0 [16.0 to 48.0] | 20.0 [6.00 to 72.1]

3. Primary Outcome: Area Under the Serum Concentration Time Curve From Time Zero to Time of Last Quantifiable Concentration (AUClast) of Efavaleukin Alfa
Description: Blood samples were collected to determine PK parameters.
Time Frame: Day 1: Pre-dose, 6, 12, & 16 hours post-dose, and days 2 (24 hours post-dose), 3, 4, 5, 6, 8, 11, 15, 22, 29 and 43
Population: PK population: all participants who received at least 1 dose of efavaleukin alfa and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Group 1: Chinese Participants - Efavaleukin Alfa (Dose Level 1) | Group 2: Chinese Participants - Efavaleukin Alfa (Dose Level 2) | Group 3: Japanese Participants -Efavaleukin Alfa (Dose Level 2) | Group 4: Caucasian Participants - Efavaleukin Alfa (Dose Level 2)
Number analyzed (Participants) | 8 | 8 | 8 | 8
hr*ng/mL | 1530 (70.0) | 2330 (38.8) | 2590 (29.0) | 2660 (44.2)

4. Primary Outcome: Area Under the Serum Concentration Time Curve From Time Zero to Infinity (AUCinf) of Efavaleukin Alfa
Description: Blood samples were collected to determine PK parameters.
Time Frame: Day 1: Pre-dose, 6, 12, & 16 hours post-dose, and days 2 (24 hours post-dose), 3, 4, 5, 6, 8, 11, 15, 22, 29 and 43
Population: PK population: all participants who received at least 1 dose of efavaleukin alfa and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Group 1: Chinese Participants - Efavaleukin Alfa (Dose Level 1) | Group 2: Chinese Participants - Efavaleukin Alfa (Dose Level 2) | Group 3: Japanese Participants -Efavaleukin Alfa (Dose Level 2) | Group 4: Caucasian Participants - Efavaleukin Alfa (Dose Level 2)
Number analyzed (Participants) | 7 | 8 | 8 | 8
hr*ng/mL | 1700 (66.7) | 2350 (38.1) | 2590 (29.0) | 2500 (43.0)

5. Secondary Outcome: Number of Participants Who Experienced One or More Treatment-emergent Adverse Events (TEAEs)
Description: Adverse events (AEs) were defined as any untoward medical occurrence in clinical study participant irrespective of a causal relationship with the study treatment. TEAEs were any event that occurred after the participant had received study treatment. Any clinically significant changes in physical examinations, clinical laboratory tests and vital signs were recorded as TEAEs.
  Serious AEs (SAEs) were defined as any event that met at least 1 of the following serious criteria:
  * Resulted in death (fatal)
  * Required in-patient hospitalization or prolongation of existing hospitalization
  * Resulted in persistent or significant disability/incapacity
  * A congenital anomaly/birth defect
  * Other medically important serious event
Time Frame: Day 1 to Day 43
Population: Safety population: all participants who received at least 1 dose of efavaleukin alfa and had at least 1 post-dose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Chinese Participants - Efavaleukin Alfa (Dose Level 1) | Group 2: Chinese Participants - Efavaleukin Alfa (Dose Level 2) | Group 3: Japanese Participants -Efavaleukin Alfa (Dose Level 2) | Group 4: Caucasian Participants - Efavaleukin Alfa (Dose Level 2)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Participants
  All TEAEs | 8 | 8 | 8 | 8
  Serious TEAEs | 1 | 0 | 1 | 0

6. Secondary Outcome: Number of Participants With Anti-Efavaleukin Alfa Antibodies and Anti-Interleukin 2 (IL-2) Antibodies
Description: Number of participants who tested positive for developing anti-efavaleukin alfa antibodies and/or anti-IL2 antibodies at 1 or more post-baseline time points, who had a negative or no result at baseline.
Time Frame: Day 1 up to Day 43
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Chinese Participants - Efavaleukin Alfa (Dose Level 1) | Group 2: Chinese Participants - Efavaleukin Alfa (Dose Level 2) | Group 3: Japanese Participants -Efavaleukin Alfa (Dose Level 2) | Group 4: Caucasian Participants - Efavaleukin Alfa (Dose Level 2)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Participants
  Anti-Efavaleukin Alfa Antibodies | 6 | 7 | 7 | 7
  Anti-IL-2 Antibodies | 0 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: Day 1 to Day 43
Description: AEs were defined as any untoward medical occurrence in clinical study participant irrespective of a causal relationship with the study treatment. TEAEs were any event that occurred after the participant had received study treatment.
Arm/Group | Group 1: Chinese Participants - Efavaleukin Alfa (Dose Level 1) | Group 2: Chinese Participants - Efavaleukin Alfa (Dose Level 2) | Group 3: Japanese Participants -Efavaleukin Alfa (Dose Level 2) | Group 4: Caucasian Participants - Efavaleukin Alfa (Dose Level 2)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/8 | 1/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 8/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Chinese Participants - Efavaleukin Alfa (Dose Level 1) (N=8) | Group 2: Chinese Participants - Efavaleukin Alfa (Dose Level 2) (N=8) | Group 3: Japanese Participants -Efavaleukin Alfa (Dose Level 2) (N=8) | Group 4: Caucasian Participants - Efavaleukin Alfa (Dose Level 2) (N=8)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Chinese Participants - Efavaleukin Alfa (Dose Level 1) (N=8) | Group 2: Chinese Participants - Efavaleukin Alfa (Dose Level 2) (N=8) | Group 3: Japanese Participants -Efavaleukin Alfa (Dose Level 2) (N=8) | Group 4: Caucasian Participants - Efavaleukin Alfa (Dose Level 2) (N=8)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site discolouration (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 6 (6) | 7 (7) | 5 (5) | 7 (7)
Injection site pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 2 (2) | 1 (1) | 4 (4) | 2 (2)
Injection site rash (General disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sars-cov-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 3 (3) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Urticaria papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/33/NCT04987333/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT04987333/SAP_001.pdf